CLINICAL TRIAL: NCT04449887
Title: The Role of Intestinal Flora in the Pathogenesis of FD and the Intervention of Xiangsha Liujunzi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ZZ13-YQ-006
Record Dates: First submitted 2020-06-06; First posted 2020-06-29 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Functional Dyspepsia
Keywords: xiangshaliujunzi,functional dyspepsia，Intestinal flora

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The treatment group (Experimental): The subjects in this group were treated with Xiangsha Liujunzi granule for 4 weeks
  Interventions: Drug: Xiangsha Liujunzi granules

INTERVENTIONS:
Drug: Xiangsha Liujunzi granules — A traditional Chinese medicine compound, taken three times a day, one bag at a time, for a total of 28 days

SUMMARY:
Functional dyspepsia (FD) is a common digestive system disease in clinic. Although it has not reached the level of life-threatening, it seriously affects the quality of life of patients. The pathogenesis of FD mainly involves gastric motility disorder and visceral hypersensitivity. At present, there are gastric motility promoting drugs and gastric acid inhibiting drugs, but they can not achieve satisfactory therapeutic effect. Traditional Chinese medicine has a good clinical effect on FD, but the specific mechanism is not clear. With the gradual deepening of intestinal flora research, it provides a useful tool for elucidating the mechanism of action of traditional Chinese medicine compound. The role of intestinal flora in the pathogenesis of FD, especially in the pathogenesis of symptoms, has not been studied, and the mechanism of Spleen-strengthening and motility-promoting effects of Xiangsha Liujun has not been studied from the perspective of intestinal flora. In this study, 16S rRNA high-throughput sequencing technology was used to observe the difference of intestinal flora between FD patients and normal people, and then to observe the effect of Xiangsha Liujun on intestinal flora of FD patients. The aim of this study was to explore the role of intestinal flora in the pathogenesis of FD and to elucidate the therapeutic mechanism of Xiangsha Liujunzi by regulating intestinal flora of FD patients, so as to provide support for follow-up clinical and experimental studies.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of functional dyspepsia by Rome IV . ② Clinical diagnosis of spleen deficiency and qi stagnation by CTM. ③ Must be able to swallow potion.

Exclusion Criteria:

* Gastric ulcer

  * Duodenal ulcer.

    * Gastroesophageal reflux disease .

      * Chronic gastritis with HP (+).

        * Chronic pancreatitis.

          * Diabetes.

            * Chronic renal insufficiency.

              * Hematological disease.

                * tumor or AIDS.

                  * Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-07-07 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
General impression scale | 4 weeks
  Significant deterioration, slight deterioration, no remission, slight remission,significant remission, complete remission.Change from baseline on different levels at 4 weeks.
Symptom severity scale | 4 weeks
  early satiety,upper abdominal pain, postprandial fullness discomfort,Burning sensation of upper abdomen.Change from baseline on symptom severity scale at 4 weeks.

SECONDARY OUTCOMES:
SF-36 scale | 4 weeks
  Eight dimensions: physiological function, social function, physiological function, physical pain, mental health, emotional function, vitality, overall health.Change from baseline on every dimension at 4 weeks.
TCM symptom score (TCMSS) | 4 weeks
  15 items: fullness of ruffles, epigastralgia, stupor, heartburn or burning sensation, belching and acid regurgitation, salivation clearing, pharyngeal obstruction, thirsty but not willing to drink water, less abdominal distention and pain, weakness of limbs, shortness of breath, laziness, heavy sleepiness of the whole body and limbs, fear of cold and cold, loose stools.Change from baseline on TCM symptom score (TCMSS) at 4 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Digestive department of Xi Yuan Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China